CLINICAL TRIAL: NCT01083693
Title: An Open Label Multicenter Post Marketing Observational Study for the Evaluation of Quality of Life Outcomes and Tolerability of HUMIRA in Routine Clinical Use in Patients With RA PsA AS After Unsustainable Response to Disease Modifying Antirheumatic Drugs and or Biologicals
Brief Title: Quality of Life Outcomes of HUMIRA in Rheumatoid Arthritis (RA), Psoriatic Arthritis (PsA), Ankylosing Spondylitis (AS) After Unsustainable Response to Biologicals and Disease Modifying Antirheumatic Drugs
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Group Data Management Biostatistics (Unknown)
Responsible Party: Dr. Astrid Dworan-Timler, Medical Director, Abbott AUSTRIA
Other Study IDs: P10-726
Record Dates: First submitted 2010-02-28; First posted 2010-03-10 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: Monoclonals; Antibodies; Ankylosing Spondylitis; Antirheumatic Agents; Quality of Life; Adalimumab; rheumatoid arthritis; psoriatic arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid, Psoriatic Arthritis, Ankylosing Spondylitis: Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, patients with unsustainable clinical response to disease modifying antirheumatic drugs and or biological disease modifying antirheumatic drugs.

SUMMARY:
The aim of this post-marketing observational study is to obtain further data on the evaluation of quality of life outcomes of HUMIRA® in routine clinical use in patients with Rheumatoid Arthritis (RA), Psoriatic Arthritis (PsA) or Ankylosing Spondylitis (AS) after unsustainable clinical response to disease modifying antirheumatic drugs (DMARD) and or biological disease modifying antirheumatic drugs (BDMARD). Treatment strategies in moderate to severe rheumatoid arthritis, psoriatic arthritis and in severe active ankylosing spondylitis commonly consist of introducing biologics after conventional disease modifying antirheumatic drugs or non steroidal antiinflammatory drugs fail. Although biologic disease modifying antirheumatic drugs are generally well-tolerated, intolerances may develop or efficacy may diminish, at which time another biologic disease modifying antirheumatic drug might be considered. This study shall evaluate the quality of life outcomes of HUMIRA®, given after conventional disease modifying antirheumatic drugs and or non antiinflammatory drug failures and or after biological disease modifying antirheumatic drug failures . Failure in this context means primary or secondary loss of efficacy or intolerance to the initial agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients age greater than or equal to 18
* Patients must fulfill international and national guidelines for use of a BDMARD in RA, PsA and AS (Chest X-ray and purified protein derivative (PPD) skin test negative for tuberculosis).

In addition one of the following criteria must be fulfilled:

* unsatisfactory DMARD response defined as failure to treatment with at least two DMARDs including Methotrexate in patients with RA or PsA
* unsatisfactory NSAID response in patients with AS or
* unsatisfactory response to prior BDMARDs (in this case patients must have received BDMARDs at least 12 weeks before visit 1) in patients with RA or PsA or AS.

Exclusion Criteria:

* Patients who meet contraindications as outlined in the latest version of the Humira syringe® Summary of Product Characteristics (SmPC) and Humira Pen® SmPC
* Patients participating in another study or clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic and medical practice specialized in rheumatology
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Dworan-Timler, MD, Study Director — Abbott AUSTRIA
Locations (20):
- Austria (20):
  - Site Reference ID/Investigator # 32372, Amstetten
  - Site Reference ID/Investigator # 32368, Bludenz
  - Site Reference ID/Investigator # 32367, Gloggnitz
  - Site Ref # / Investigator 37123, Graz
  - Site Ref # / Investigator 37125, Innsbruck
  - Site Reference ID/Investigator # 32375, Klagenfurt
  - Site Reference ID/Investigator # 32365, Linz
  - Site Reference ID/Investigator # 32369, Linz
  - Site Reference ID/Investigator # 32371, Linz
  - Site Reference ID/Investigator # 32376, Linz
  - Site Reference ID/Investigator # 32373, Neudorf
  - Site Reference ID/Investigator # 32364, Salzburg
  - Site Reference ID/Investigator # 18782, Vienna
  - Site Reference ID/Investigator # 32363, Vienna
  - Site Reference ID/Investigator # 32377, Vienna
  - Site Reference ID/Investigator # 32378, Vienna
  - Site Reference ID/Investigator # 32366, Vienna
  - Site Reference ID/Investigator # 32374, Vöcklabruck
  - Site Reference ID/Investigator # 32370, Weiz
  - Site Ref # / Investigator 37124, Wels

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 162 participants were screened for this study. Of those, 161 are included in the analysis as one participant was a screen failure.
Groups:
- Rheumatoid Arthritis (RA): Rheumatoid Arthritis participants with unsustainable clinical response to disease modifying antirheumatic drugs and or biological disease modifying antirheumatic drugs.
- Psoriasis Arthritis (PsA): Psoriatic Arthritic participants with unsustainable clinical response to disease modifying antirheumatic drugs and or biological disease modifying antirheumatic drugs.
- Ankylosing Spondylitis (AS): Ankylosing Spondylitis participants with unsustainable clinical response to nonsteroidal antiinflammatory drugs and or biological disease modifying antirheumatic drugs.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Ankylosing Spondylitis (AS)
Started | 93 | 28 | 40
Completed | 73 | 22 | 33
Not Completed | 20 | 6 | 7
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Lack of effectiveness | 13 | 2 | 2
Not completed — Patient Moved | 0 | 1 | 0
Not completed — Complete remission | 0 | 1 | 0
Not completed — Other medical condition/surgery | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 2
Not completed — Reason unknown | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Ankylosing Spondylitis (AS) | Total
Number analyzed (Participants) | 93 | 28 | 40 | 161
Age Continuous [Mean (Standard Deviation); unit: years] | 55.7 (14.2) | 47.9 (8.1) | 42.0 (12.9) | 50.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 9 | 17 | 101
  Male | 18 | 19 | 23 | 60
Region of Enrollment [Number; unit: participants]
  Austria | 93 | 28 | 40 | 161
Duration of underlying disease [Mean (Standard Deviation); unit: years] — Average duration (years) of underlying disease
  years | 7.6 (7.4) | 6.2 (6.8) | 8.9 (11.4) | 7.7 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: RA and if Reasonable for PsA Patients Health Assessment Questionnaire Disability Index HAQ-DI
Description: The HAQ-DI is a questionnaire that measures functional status (disability) and health-related quality of life. It measures a patient's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene,reach, grip, activities. Each question is evaluated according to the degree of severity on a scale ranging from 0 (without any difficulty) to 3 (unable to do).
Time Frame: Baseline, months 3,6,9,12
Population: Mean (average) score is based on the number of participants included in the analysis (N =121) who completed the assessment at each timepoint (Baseline, 3, 6, 9 and 12 months and early termination [for participants who discontinued the study early]) in each disease group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Total
Number analyzed (Participants) | 93 | 28 | 121
Units on a scale
  Baseline | 1.2 (0.7) | 0.9 (0.7) | 1.1 (0.7)
  3 months | 0.9 (0.7) | 0.4 (0.4) | 0.8 (0.7)
  6 months | 0.8 (0.6) | 0.4 (0.5) | 0.7 (0.6)
  9 months | 0.8 (0.6) | 0.3 (0.5) | 0.7 (0.6)
  12 months | 0.7 (0.6) | 0.2 (0.3) | 0.6 (0.6)
  Early Termination | 1.4 (0.9) | 0.0 (0.0) | 1.2 (1.0)

2. Primary Outcome: SF-36 as Generic Measure of Health Status for RA, PsA, AS Physical Score Measures How Decrements in Physical Function Affect Day-to-day Activities Impact of Physical Impairment/Disability on QoL ,Mental Score: Impact of Mental Effect, Symptoms of Pain
Description: Medical Outcomes Study Short Form 36 (MOS SF-36) is generic assessment of health status that consists of 36 questions within 8 domains including Physical Functioning (PF), Role Functioning - Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Functioning - Emotional (RE), Mental Health (MH) and Reported Health Transition (HT). Results from each domain are summarized and transformed into a scale ranging from 0 (worst) to 100 (best) with the exception of HT. The score range for HT is 0 (worst) to 5 (best).
Time Frame: Baseline, months 3,6,9,12
Population: Mean (average) score is based on the number of participants included in the analysis (N=161) who completed the assessment at each timepoint (Baseline, 3, 6, 9 and 12 months and early termination [participants who discontinued the study early]) in each disease group. No participants in the PsA or the AS group attended an early termination visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Ankylosing Spondylitis (AS) | Total
Number analyzed (Participants) | 93 | 28 | 40 | 161
Units on a scale
  Physical Functioning -Baseline | 51.4 (26.4) | 58.1 (26.2) | 53.3 (23.4) | 53.1 (25.6)
  Physical Functioning - 3 months | 67.4 (24.3) | 74.3 (21.3) | 76.5 (21.9) | 71.0 (23.4)
  Physical Functioning - 6 months | 65.3 (24.4) | 76.0 (21.9) | 79.4 (22.2) | 70.9 (24.1)
  Physical Functioning - 9 months | 67.4 (24.6) | 79.8 (19.5) | 81.4 (18.7) | 73.4 (23.1)
  Physical Functioning -12 months | 70.3 (23.8) | 85.9 (13.2) | 80.4 (24.5) | 75.9 (23.1)
  Physical Functioning - Early Termination | 33.3 (28.6) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 33.3 (28.6)
  Role Functioning -Physical - Baseline | 29.8 (40.5) | 38.9 (43.5) | 25.0 (32.2) | 30.3 (39.2)
  Role Functioning - Physical - 3 months | 57.3 (43.5) | 58.7 (41.0) | 67.4 (38.8) | 60.2 (41.8)
  Role Functioning - Physical - 6 months | 55.3 (44.0) | 70.2 (36.8) | 73.4 (37.6) | 62.7 (41.7)
  Role Functioning - Physical - 9 months | 55.4 (43.7) | 72.5 (40.5) | 75.0 (37.2) | 63.8 (42.1)
  Role Functioning - Physical - 12 months | 59.8 (42.3) | 85.0 (28.6) | 75.9 (38.9) | 68.9 (40.1)
  Role Functioning - Physical - Early Termination | 29.2 (40.1) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 29.2 (40.1)
  Bodily Pain - Baseline | 33.6 (19.2) | 36.6 (23.9) | 27.7 (19.1) | 32.7 (20.2)
  Bodily Pain- 3 months | 56.5 (24.3) | 61.0 (23.5) | 66.1 (24.9) | 59.8 (24.5)
  Bodily Pain- 6 months | 53.9 (19.9) | 64.9 (23.7) | 67.7 (25.2) | 59.5 (22.8)
  Bodily Pain- 9 months | 59.5 (21.6) | 69.3 (25.9) | 69.8 (22.5) | 64.0 (23.0)
  Bodily Pain- 12 months | 62.5 (19.1) | 74.0 (23.2) | 71.2 (27.9) | 67.0 (22.8)
  Bodily Pain- Early Termination | 25.7 (37.6) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 25.7 (37.6)
  General Health - Baseline | 42.9 (19.4) | 41.9 (18.9) | 39.1 (16.4) | 41.8 (18.6)
  General Health - 3 months | 51.7 (17.9) | 53.0 (20.8) | 59.0 (21.7) | 53.8 (19.5)
  General Health - 6 months | 54.0 (16.6) | 61.6 (18.0) | 60.1 (23.7) | 57.0 (19.1)
  General Health - 9 months | 54.9 (19.0) | 59.8 (19.1) | 65.7 (22.1) | 58.7 (20.3)
  General Health - 12 months | 59.5 (20.2) | 65.0 (18.1) | 66.3 (23.0) | 62.3 (20.7)
  General Health - Early Termination | 39.0 (26.2) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 39.0 (26.2)
  Vitality - Baseline | 39.3 (19.0) | 39.8 (21.1) | 32.4 (18.7) | 37.7 (19.5)
  Vitality - 3 months | 53.6 (19.3) | 53.3 (19.7) | 54.5 (20.4) | 53.8 (19.5)
  Vitality - 6 months | 52.6 (16.0) | 56.8 (19.4) | 57.9 (19.4) | 54.7 (17.5)
  Vitality - 9 months | 52.3 (19.1) | 56.3 (16.0) | 59.2 (20.1) | 54.9 (19.0)
  Vitality - 12 months | 56.9 (17.7) | 65.0 (14.9) | 58.0 (21.5) | 58.7 (18.4)
  Vitality - Early Termination | 23.3 (16.3) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 23.3 (16.3)
  Social Functioning - Baseline | 59.5 (30.0) | 66.2 (31.2) | 52.8 (25.0) | 59.1 (29.2)
  Social Functioning - 3 months | 75.3 (20.9) | 79.3 (18.7) | 78.0 (21.4) | 76.8 (20.6)
  Social Functioning - 6 months | 78.4 (20.5) | 85.7 (19.1) | 81.0 (23.0) | 80.4 (21.0)
  Social Functioning - 9 months | 79.0 (19.7) | 86.9 (20.1) | 83.2 (23.2) | 81.5 (20.8)
  Social Functioning - 12 months | 82.3 (20.4) | 93.1 (14.3) | 80.4 (25.1) | 83.8 (21.1)
  Social Functioning - Early Termination | 47.9 (31.0) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 47.9 (31.0)
  Role Functioning -Emotional - Baseline | 45.1 (44.7) | 55.6 (43.4) | 40.7 (42.2) | 46.0 (43.8)
  Role Functioning -Emotional - 3 months | 66.2 (42.3) | 75.4 (41.7) | 74.0 (35.7) | 69.8 (40.5)
  Role Functioning -Emotional - 6 months | 69.7 (41.2) | 82.5 (35.9) | 76.3 (36.7) | 73.7 (39.2)
  Role Functioning -Emotional - 9 months | 72.4 (40.5) | 78.3 (39.4) | 81.6 (31.6) | 76.0 (38.0)
  Role Functioning -Emotional - 12 months | 78.2 (37.0) | 91.7 (26.2) | 75.0 (38.1) | 79.9 (35.7)
  Role Functioning - Emotional - Early Termination | 33.3 (51.6) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 33.3 (51.6)
  Mental Health - Baseline | 55.6 (21.5) | 63.1 (22.1) | 53.9 (21.0) | 56.6 (21.6)
  Mental Health - 3 months | 66.1 (18.8) | 70.1 (19.0) | 70.4 (18.9) | 67.9 (18.9)
  Mental Health - 6 months | 67.9 (16.3) | 75.8 (16.6) | 73.6 (18.9) | 70.8 (17.3)
  Mental Health - 9 months | 70.7 (17.5) | 74.6 (21.1) | 76.1 (18.8) | 72.9 (18.6)
  Mental Health - 12 months | 73.2 (14.8) | 81.8 (13.9) | 76.7 (17.2) | 75.8 (15.5)
  Mental Health - Early Termination | 41.3 (23.8) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 41.3 (23.8)
  Reported Health Transition - Baseline | 3.5 (1.2) | 3.5 (1.1) | 3.9 (1.1) | 3.6 (1.2)
  Reported Health Transition - 3 months | 2.0 (1.1) | 2.1 (1.1) | 1.8 (1.1) | 2.0 (1.1)
  Reported Health Transition - 6 months | 2.1 (1.0) | 1.8 (1.0) | 1.5 (0.8) | 1.9 (1.0)
  Reported Health Transition - 9 months | 1.9 (0.8) | 1.8 (1.0) | 1.4 (0.6) | 1.7 (0.8)
  Reported Health Transition - 12 months | 1.7 (0.9) | 1.4 (0.6) | 1.7 (0.9) | 1.6 (0.9)
  Reported Health Transition - Early Termination | 3.5 (2.0) | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | NA (NA) — Score not available as there were no participants who had an early termination visit in this group. | 3.5 (2.0)

3. Primary Outcome: EQ-5D for RA,PsA,AS, as Measure of Health Outcome. Self Reported Health Status: Measures Mobility, Self Care, Usual Activities, Pain Discomfort, Anxiety Depression
Description: European Quality of Life 5 Dimensions (EQ-5D) is a self-reported health outcome which measures mobility, self care, usual activities, pain discomfort, anxiety depression. An overall score is derived that measures from -0.59 (worst) to +1 (best).
  In addition, health state is measured on the thermometer scale (score 0 to 100) with higher scores representing better health status.
Time Frame: Baseline, months 3,6,9,12
Population: Mean (average) score is based on the number of participants included in the analysis (N=161) who completed the assessment at each timepoint (Baseline, 3, 6, 9 and 12 months and early termination [for participants who discontinued the study early]) in each disease group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Ankylosing Spondylitis (AS) | Total
Number analyzed (Participants) | 93 | 28 | 40 | 161
Units on a scale
  EQ-5D - Baseline | 0.5 (0.3) | 0.5 (0.3) | 0.4 (0.3) | 0.5 (0.3)
  EQ-5D - 3 months | 0.7 (0.2) | 0.8 (0.2) | 0.8 (0.2) | 0.7 (0.2)
  EQ-5D - 6 months | 0.7 (0.2) | 0.8 (0.1) | 0.8 (0.3) | 0.8 (0.2)
  EQ-5D - 9 months | 0.7 (0.2) | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2)
  EQ-5D - 12 months | 0.8 (0.2) | 0.8 (0.1) | 0.8 (0.3) | 0.8 (0.2)
  EQ-5D - Early Termination | 0.3 (0.5) | 1.0 (NA) — Only one patient completed this assessment at an early termination visit therefore a standard deviation value is not available. | NA (NA) — There were no patients who completed this assessment at an early termination visit in this group/arm. | 0.4 (0.5)
  Thermometer Scale - Baseline | 49.0 (21.5) | 52.5 (24.8) | 40.2 (22.6) | 47.4 (22.7)
  Thermometer Scale - 3 months | 64.8 (22.0) | 68.7 (21.0) | 64.9 (25.6) | 65.5 (22.7)
  Thermometer Scale - 6 months | 59.5 (22.0) | 68.9 (23.3) | 68.7 (29.0) | 63.7 (24.5)
  Thermometer Scale - 9 months | 67.5 (21.0) | 67.8 (25.2) | 69.2 (25.0) | 68.0 (22.8)
  Thermometer Scale - 12 months | 73.2 (18.5) | 79.2 (16.0) | 71.5 (28.5) | 73.9 (21.2)
  Thermometer Scale - Early Termination | 67.2 (29.1) | 100.0 (NA) — Only one patient completed this assessment at an early termination visit therefore a standard deviation value is not available. | NA (NA) — There were no patients who completed this assessment at an early termination visit in this group/arm. | 71.9 (29.3)

4. Secondary Outcome: DAS28: Changes in Disease Activity Score 28 in Patients With RA and if Reasonable in PsA: Measures the no. of Swollen and Tender Joints (28 Joints), Erythrocyte Sedimentation Rate, Patients Global Assessment of Disease Activity on a Visual Scale
Description: The Disease Activity Score 28 measures disease activity based on the number of swollen and tender joints (28 joints), erythrocyte sedimentation rate, and patient's global assessment of disease activity on a visual scale. DAS28 is a unit scale from 0 (best value) to 10.0 (worst value).
Time Frame: Baseline,months 3,6,9,12
Population: Mean (average) score is based on the number of participants included in the analysis (N=121) who completed the assessment at each timepoint (Baseline, 3, 6, 9 and 12 months and early termination [for participants who discontinued the study early]) in each disease group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Total
Number analyzed (Participants) | 93 | 28 | 121
Units on a scale
  Baseline | 5.4 (1.2) | 4.9 (1.1) | 5.3 (1.2)
  3 months | 3.8 (1.5) | 3.0 (1.1) | 3.7 (1.5)
  6 months | 3.4 (1.2) | 2.4 (1.0) | 3.2 (1.2)
  9 months | 3.7 (1.5) | 2.5 (1.0) | 3.4 (1.5)
  12 months | 3.4 (1.3) | 2.5 (1.0) | 3.2 (1.3)
  Early Termination | 5.3 (1.8) | 2.1 (0.8) | 4.5 (2.2)

5. Secondary Outcome: Changes in Bath Ankylosing Spondylitis Disease Activity Index in Patients With AS: Measures Patients Fatigue, Pain (Neck, Hip, Other Joints), Tender Sensitive Body Sites, Morning Stiffness
Description: Bath as Disease Activity Index (BASDI) measures fatigue, pain (neck, hip, other joints), tender sensitive body sites, and morning stiffness for patients suffering from AS. Scores range from 0 to 10 with higher scores representing worse disease activity.
Time Frame: Baseline, months 3,6,9,12
Population: Mean (average) score is based on the number of participants included in the analysis (N=40) who completed the assessment at each timepoint (Baseline, 3, 6, 9 and 12 months and early termination [for participants who discontinued the study early]).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ankylosing Spondylitis (AS)
Number analyzed (Participants) | 40
Units on a scale
  Baseline | 6.0 (1.6)
  3 months | 2.8 (2.1)
  6 months | 2.0 (1.5)
  9 months | 2.4 (2.0)
  12 months | 2.5 (2.3)
  Early Termination | 4.6 (3.3)

6. Secondary Outcome: Physician´s /Patient's Global Assessment on Disease Activity Measured on a Visual Analogue Scale, for RA and PsA Patients Only
Description: Physician's and Patient's Global Assessment of Disease Activity (PGA) are measured using a visual analogue scale with scores ranging from 0 to 100 (higher scores indicate worse disease activity).
Time Frame: Baseline, months 3,6,9,12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Total
Number analyzed (Participants) | 93 | 28 | 121
Units on a scale
  Physician's PGA - Baseline | 55.1 (19.6) | 52.0 (26.9) | 54.4 (21.4)
  Physician's PGA - 3 months | 28.8 (21.1) | 29.0 (20.1) | 28.9 (20.8)
  Physician's PGA - 6 months | 29.5 (20.2) | 23.1 (19.7) | 28.1 (20.2)
  Physician's PGA - 9 months | 28.6 (19.5) | 17.9 (13.1) | 26.1 (18.7)
  Physician's PGA - 12 months | 22.9 (16.8) | 19.4 (14.7) | 22.1 (16.3)
  Physician's PGA - Early Termination | 57.0 (30.5) | 11.7 (12.6) | 47.3 (33.4)
  Patient's PGA - Baseline | 60.0 (23.3) | 58.3 (27.6) | 59.6 (24.3)
  Patient's PGA - 3 months | 32.4 (22.9) | 34.3 (22.3) | 32.8 (22.7)
  Patient's PGA - 6 months | 32.1 (21.1) | 27.7 (21.9) | 31.1 (21.2)
  Patient's PGA - 9 months | 32.2 (21.1) | 22.0 (16.9) | 29.9 (20.6)
  Patient's PGA - 12 months | 26.1 (18.4) | 23.9 (15.9) | 25.6 (17.8)
  Patient's PGA - Early Termination | 63.2 (29.5) | 21.7 (29.3) | 54.9 (33.2)

7. Secondary Outcome: Physician´s / Patient's Global Assessment of State of Health (GH) Measured on a Visual Analogue Scale, for RA and PsA Patients Only
Description: Physician's and Patient's Global Assessment of State of Health was measured using a visual analogue scale with scores from 0 to 100 (higher scores indicate worse health state).
Time Frame: Baseline, months 3,6,9,12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Total
Number analyzed (Participants) | 93 | 28 | 121
Units on a scale
  Physician's GH - Baseline | 51.4 (21.0) | 46.8 (23.7) | 50.4 (21.6)
  Physician's GH -3 months | 29.9 (22.3) | 25.3 (19.3) | 28.9 (21.6)
  Physician's GH - 6 months | 31.5 (21.4) | 26.2 (23.9) | 30.4 (21.9)
  Physician's GH - 9 months | 31.3 (22.4) | 26.5 (24.5) | 30.2 (22.8)
  Physician's GH - 12 months | 29.0 (24.1) | 26.2 (26.7) | 28.3 (24.6)
  Physician's GH - Early Termination | 56.2 (28.6) | 11.7 (12.6) | 46.6 (31.8)
  Patient's GH - Baseline | 55.3 (25.4) | 59.0 (24.8) | 56.1 (25.2)
  Patient's GH -3 months | 33.6 (23.2) | 31.4 (23.4) | 33.1 (23.2)
  Patient's GH - 6 months | 32.9 (22.3) | 29.4 (26.6) | 32.1 (23.2)
  Patient's GH -9 months | 35.0 (22.7) | 26.9 (23.4) | 33.2 (23.0)
  Patient's GH -12 months | 30.4 (23.7) | 30.6 (25.7) | 30.4 (24.0)
  Patient's GH - Early Termination | 62.5 (32.1) | 21.7 (29.3) | 53.8 (35.0)

8. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: Erythrocyte sedimentation rate (ESR) is a nonspecific lab value that measures inflammation from arthritic disease. A decrease in the level indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, months 3,6,9,12
Population: Mean (average) value is based on the number of participants included in the analysis (N=161) who completed the lab assessment at each timepoint (Baseline, 3, 6, 9 and 12 months and early termination [for participants who discontinued the study early]) in each disease group.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Ankylosing Spondylitis (AS) | Total
Number analyzed (Participants) | 93 | 28 | 40 | 161
milligrams per deciliter (mg/dL)
  Baseline | 35.8 (22.9) | 31.7 (19.9) | 25.2 (15.7) | 32.4 (21.2)
  3 months | 25.3 (20.8) | 16.0 (13.9) | 12.4 (12.3) | 20.6 (18.8)
  6 months | 23.9 (21.9) | 12.3 (13.6) | 11.9 (10.2) | 19.0 (19.2)
  9 months | 24.2 (22.8) | 11.6 (10.2) | 11.9 (8.4) | 19.1 (19.4)
  12 months | 18.3 (13.4) | 10.5 (7.7) | 14.0 (12.8) | 15.9 (12.7)
  Early termination | 47.3 (29.1) | 18.0 (26.5) | 10.5 (2.1) | 37.3 (30.5)

9. Secondary Outcome: C-Reactive Protein
Description: The test for C-Reactive Protein (CRP) is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, months 3,6,9,12
Population: Mean (average) value is based on the number of participants included in the analysis (N =161) who completed the lab assessment at each timepoint (Baseline, 3, 6, 9 and 12 months and early termination [for participants who discontinued the study early]) in each disease group.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Ankylosing Spondylitis (AS) | Total
Number analyzed (Participants) | 93 | 28 | 40 | 161
milligrams per deciliter (mg/dL)
  Baseline | 1.9 (2.5) | 1.1 (1.0) | 1.4 (1.4) | 1.7 (2.1)
  3 months | 1.2 (2.5) | 0.7 (1.4) | 0.5 (0.6) | 0.9 (2.0)
  6 months | 1.0 (2.2) | 0.4 (1.0) | 0.4 (0.6) | 0.8 (1.8)
  9 months | 1.0 (2.6) | 0.2 (0.2) | 0.4 (0.3) | 0.7 (2.1)
  12 months | 0.4 (0.4) | 0.2 (0.2) | 0.7 (1.6) | 0.4 (0.9)
  Early Termination | 3.5 (4.7) | 1.1 (2.1) | 0.4 (0.3) | 2.6 (4.1)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected throughout the study (12 months) and 70 days following the last dose of adalimumab.
Description: A total of 15 out of 161 participants had at least one adverse event. Percentages for individual adverse events are calculated for each disease group (based on the number of participants in each group) as well as the total number of participants overall.
Arm/Group | Rheumatoid Arthritis (RA) | Psoriasis Arthritis (PsA) | Ankylosing Spondylitis (AS) | Total
Serious Adverse Events (participants affected / at risk) | 6/93 | 2/28 | 0/40 | 8/161
Other Adverse Events (participants affected / at risk) | 10/93 | 1/28 | 1/40 | 12/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis (RA) (N=93) | Psoriasis Arthritis (PsA) (N=28) | Ankylosing Spondylitis (AS) (N=40) | Total (N=161)
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Ulcer (General disorders) | 1 | 0 | 0 | 1
Arthroscopy (Investigations) | 1 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Leg amputation (Surgical and medical procedures) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis (RA) (N=93) | Psoriasis Arthritis (PsA) (N=28) | Ankylosing Spondylitis (AS) (N=40) | Total (N=161)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Uriticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Synovectomy (Surgical and medical procedures) | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.